CLINICAL TRIAL: NCT04311424
Title: Disposition of [14C]-Tirzepatide Following Subcutaneous Administration in Healthy Male Subjects
Brief Title: Study of Tirzepatide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 17378; I8F-MC-GPHX (Other: Eli Lilly and Company); 2019-003664-44 (EudraCT Number)
Record Dates: First submitted 2020-03-16; First posted 2020-03-17 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 14C Tirzepatide (Experimental): A single dose of [14C]-tirzepatide administered subcutaneously (SC).
  Interventions: Drug: 14C Tirzepatide

INTERVENTIONS:
Drug: 14C Tirzepatide — Administered SC.
  Other Names: LY3298176

SUMMARY:
The purpose of this study is to look at how much tirzepatide gets into the bloodstream and how long the body takes to get rid of it. This study will involve a single dose of 14C radiolabelled tirzepatide. This means that a radioactive tracer substance, C14, will be incorporated into the study drug to investigate the study drug and its breakdown products and to find out how much of these pass from blood into urine, feces and expired air.

Screening is required within 28 days prior to the start of the study. For each participant, the total duration of the clinical trial will be approximately 15 weeks, including screening.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males as determined by medical history, physical examination, and other screening procedures
* Have a body mass index (BMI) between 18.0 to 32.0 kilograms per meter squared (kg/m²), inclusive at screening
* Are willing to be available for the full duration of the study

Exclusion Criteria:

* Have known allergies to tirzepatide or related compounds
* Have a medical condition or medical history that makes participation in the study unsafe or which may interfere in the interpretation of the results of the study
* Have had exposure to significant radiation within 12 months prior to dosing (for example, multiple x-ray or computed tomography [CT] scans, barium meal, being employed in a job requiring radiation exposure monitoring)
* Have participated in any clinical trial involving a radiolabeled substance within the past 12 months

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2020-10-02 (Actual); Study Completion 2020-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Ltd, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- [14C]-Tirzepatide: Participants received single dose of approximately 4.1 milligrams (mg) tirzepatide containing approximately 100 microcurie (μCi) of [14C]- tirzepatide administered as a subcutaneous injection.
Period: Overall Study
Arm/Group | [14C]-Tirzepatide
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- [14C]-Tirzepatide: Participants received single dose of approximately 4.1 mg tirzepatide containing approximately 100 μCi of [14C]- tirzepatide administered as a subcutaneous injection.
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 6

OUTCOME MEASURES:

1. Primary Outcome: Urinary Excretion of Tirzepatide Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered
Description: Urinary Excretion of Tirzepatide Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered.
Time Frame: Pre-dose and up to 63 days post-dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage of the total radioactive dose
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
Percentage of the total radioactive dose | 49.56 (2.58)

2. Primary Outcome: Fecal Excretion of Tirzepatide Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered
Description: Fecal Excretion of Tirzepatide Radioactivity Over Time Expressed As A Percentage of the Total Radioactive Dose Administered.
Time Frame: Pre-dose and up to 63 days post-dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage of the total radioactive dose
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
Percentage of the total radioactive dose | 20.46 (2.05)

3. Secondary Outcome: Total Number of Metabolites
Description: Total Number of Metabolites.
Time Frame: Pre-dose and up to 63 days post-dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Number; unit: metabolites
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
metabolites
  Plasma | 4
  Urine | 6
  Feces | 6

4. Secondary Outcome: Total Radioactivity Recovered in Urine, Feces, and Expired Air (if Applicable)
Description: Total Radioactivity Recovered in Urine, Feces, and Expired Air (if Applicable).
Time Frame: Pre-dose and up to 63 days post-dose
Population: All randomized participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage of the total radioactive dose
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
Percentage of the total radioactive dose | 70.03 (1.98)

5. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Zero To Infinity (AUC[0-∞]) of Tirzepatide
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Zero To Infinity (AUC[0-∞]) of tirzepatide.
Time Frame: Pre-dose, Day 1, 2, 3, 4, 5, 6, 7, 10, 12, 14, 22, 29, 36, 43, 50, 57, and 64 post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data of tirzepatide.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
nanogram*hour per milliliter (ng*h/mL) | 96100 (13)

6. Secondary Outcome: PK: Maximum Concentration (Cmax) of Tirzepatide
Description: PK: Maximum Concentration (Cmax) of tirzepatide.
Time Frame: Pre-dose, Day 1, 2, 3, 4, 5, 6, 7, 10, 12, 14, 22, 29, 36, 43, 50, 57, and 64 post dose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data of tirzepatide.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
ng/mL | 453 (29)

7. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Zero To Infinity (AUC[0-∞]) of Total Radioactivity
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve (AUC) From Zero To Infinity (AUC[0-∞]) of Total Radioactivity. Total radioactivity is reported as hours*nanogram equivalents per milliliter (h*ng Eq/mL).
Time Frame: Pre-dose, Day 1, 2, 3, 4, 5, 6, 7, 10, 12, 14, 22, 29, 36, 43, 50, 57, and 64 post dose
Population: All randomized participants who received at least one dose and had evaluable PK data for total radioactivity.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng Eq/mL
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
h*ng Eq/mL
  Plasma | 87900 (13)
  Whole blood | 44000 (11)

8. Secondary Outcome: PK: Maximum Concentration (Cmax) of Total Radioactivity
Description: PK: Cmax of total radioactivity in plasma and whole blood. The Cmax of total radioactivity in plasma and whole blood are reported as nanogram equivalents per milliliter (ng Eq/mL).
Time Frame: Pre-dose, Day 1, 2, 3, 4, 5, 6, 7, 10, 12, 14, 22, 29, 36, 43, 50, 57, and 64 post dose
Population: All randomized participants who received at least one dose and had evaluable PK data for total radioactivity.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng Eq/mL
Arm/Group | [14C]-Tirzepatide
Number analyzed (Participants) | 6
ng Eq/mL
  Plasma | 327 (16)
  Whole Blood | 173 (14)

ADVERSE EVENTS:
Time Frame: Up To Day 64
Description: All randomized participants
Arm/Group | [14C]-Tirzepatide
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | [14C]-Tirzepatide (N=6)
Palpitations (Cardiac disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Feeling of body temperature change (General disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 6 (6)
Presyncope (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-05-19): https://cdn.clinicaltrials.gov/large-docs/24/NCT04311424/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT04311424/SAP_001.pdf